CLINICAL TRIAL: NCT03929861
Title: An Open-label, Randomized, Two-treatment, Two-period, Two-sequence, Cross-over, Mono-center Bioequivalence Study to Compare Single Doses of Fluconazole 150 mg Capsule (Test Product) With Diflucan™ Capsule 150 mg (Reference) in Healthy Volunteers
Brief Title: Bioequivalence Trial to Prove Equal Blood Concentrations of Two Different Fluconazole Formulations
Acronym: Orca
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 16165; 2011-006159-13 (EudraCT Number)
Record Dates: First submitted 2019-04-17; First posted 2019-04-29 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Pharmacology, Clinical
Keywords: Fluconazole; bioequivalence; capsule
MeSH Terms: interventions — Fluconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluconazole, period 1 (Experimental): Subjects were randomized to receive a single dose of 150 mg fluconazole on Day 1 of period 1 after an overnight fast of at least 10 hours
  Interventions: Drug: Fluconazole (BAYT006267) 150 mg capsules; Drug: Fluconazole 150 mg capsules (DiflucanTM)
- Fluconazole, period 2 (Experimental): Subjects were randomized to receive a single dose of 150 mg fluconazole on Day 1 of period 2 after an overnight fast of at least 10 hours
  Interventions: Drug: Fluconazole (BAYT006267) 150 mg capsules; Drug: Fluconazole 150 mg capsules (DiflucanTM)

INTERVENTIONS:
Drug: Fluconazole (BAYT006267) 150 mg capsules — Fluconazole 150 mg
Drug: Fluconazole 150 mg capsules (DiflucanTM) — Fluconazole 150 mg

SUMMARY:
Primary Objective: To compare the bioavailability of a single dose of fluconazole 150 mg capsules (Test product) with the bioavailability of a single dose of Diflucan™ capsules, 150 mg (Reference) administered under fasting conditions in order to assess bioequivalence Secondary Objectives: To assess safety and tolerability in form of adverse events and clinical parameters (systolic/diastolic blood pressure, pulse rate, body temperature, physical examination, electrocardiogram, clinical laboratory testing, and overall tolerability) and to assess further pharmacokinetic parameters of fluconazole

DETAILED DESCRIPTION:
Clinical pharmacology

ELIGIBILITY:
Inclusion Criteria:

* Healthy males in the age between 18 and 50 years
* Subjects with a body weight of at least 50 kg and a BMI between 18.5 and 30.0 kg/m2
* Subjects had to be willing to use an acceptable method of contraception (double barrier) during the study and 2 weeks after the end of the study
* All subjects had to give their written informed consent prior to admission to the trial
* Legal capacity and subject ability to understand the nature, scope and risk/benefit of the trial

Exclusion Criteria:

* Any finding of physical examination (including blood pressure, pulse rate, and ECG) deviating from normal and of clinical relevance
* Positive test for hepatitis B surface antigen test, anti hepatitis C virus (anti-HCV), or human immunodeficiency virus (HIV)-1/2 antibodies and HIV-1 p24-antigen
* Positive drug screen test (verified by "Mahsan-Kombi/DOA2" and "Kombi 4/O2TSchnelltest"), or any history or suspicion of barbiturate, amphetamine, benzodiazepine, cocaine, opiates, and cannabis abuse
* More than moderate alcohol consumption (>40 g of alcohol regularly per day)
* Demonstrated excess in xanthine consumption (more than 5 cups of coffee or equivalent per day)
* Subjects with known hypersensitivity to fluconazole and any other excipient of the test products and subjects with lactose intolerance
* Subjects with known hypersensitivity to other azoles
* Any need of medication during the trial except allowed medication (paracetamol up to 1 g a day)
* Any concomitant medication, including herbal remedies, within 10 days before administration of the investigational medicinal product (IMP), or within a period shorter than 10 times the elimination half-life of the respective medication
* History of severe allergies, non-allergic drug reactions, multiple drug allergies or active hay fever
* Any active disease, acute or chronic
* Febrile or infectious illness within 1 week before screening
* Any other disease or condition which could influence the metabolism of the drug (e.g., endocrine diseases)
* Any gastrointestinal complaints within 1 week before screening (gastrointestinal disorders including irritable bowel and gastrointestinal ulcer)
* Any relevant history of chronic or recurrent metabolic, renal, hepatic, pulmonary, gastrointestinal (especially history of chronic gastritis or peptic ulcers), neurological (especially history of epileptic seizures), endocrinological, immunological, psychiatric or cardiovascular disease, myopathies and bleeding disorders
* Subjects with QTc intervals of more than 450 ms calculated by Bazett's formula
* Subjects with a pulse rate below 50 or above 90 beats per minute
* Subjects with serum creatinine concentrations outside the range of <1.20 mg/dL
* Subjects with a medical disorder, condition or history of such that could impair the subject's ability to participate or complete this trial in the opinion of the Investigator
* Participated in the treatment phase of another clinical trial within 30 days prior to first administration of the IMP
* Blood donation or blood sample collection exceeding 200 mL within the last 30 days
* Unwilling or unable to comply with all requirements outlined in the protocol
* Excessive sports or sauna within 5 days before start of the treatment phase
* Consumption of xanthine- and quinine-containing food and beverages and certain fruit juices such as grapefruit juice within 72 h before IMP administration
* Alcohol consumption within 24 h before screening and within 72 h before IMP administration (on Day -1 verified by alcohol breath test)
* History of alcohol or drug abuse within the last 5 years
* History of smoking (within the last 12 months before screening)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2012-07-31 (Actual); Primary Completion 2012-09-10 (Actual); Study Completion 2012-09-10 (Actual)

PRIMARY OUTCOMES:
Cmax | Pre-dose and up to 72 hours post-dose
  Concentration maximum
AUC0-tlast | Pre-dose and up to 72 hours post-dose
  Area under the plasma concentration time curve from time 0 to the last data point above the lower limit of quantification

SECONDARY OUTCOMES:
Number of participants with Adverse Events as a Measure of safety and tolerability | Up to 7 weeks
tmax | Pre-dose and up to 72 hours post-dose
  Time of maximum concentration
t½λz | Pre-dose and up to 72 hours post-dose
  Half-life associated with the terminal slope
MRT | Pre-dose and up to 72 hours post-dose
  Mean residence time

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Mannheim, Baden-Wurttemberg, Germany

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/